CLINICAL TRIAL: NCT06579274
Title: A Randomized, Placebo-controlled, Double-blind Clinical Trial Evaluating the Safety and Efficacy of Parecoxib in Hospitalized Patients With Spontaneous Subarachnoid Hemorrhage
Brief Title: Evaluation of the Safety and Efficacy of Parecoxib in Patients With Subarachnoid Hemorrhage
Acronym: PARISAH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Collaborators: Masaryk University (Other); CZECRIN - Czech Clinical Research Infrastructure Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAR-FNUSA-2024
Record Dates: First submitted 2024-08-19; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Neurological Complication
Keywords: subarachnoidal hemorrhage; inflammation; NSAIDs
MeSH Terms: conditions — Inflammation | interventions — parecoxib

STUDY DESIGN:
Intervention Model Description: The clinical trial is planned as a multicenter, prospective, randomized, double-blind, placebo-controlled Phase II clinical trial, a so-called therapeutic exploratory study. This is an investigator-initiated, academic clinical trial to evaluate the safety and efficacy of parecoxib in hospitalized patients with spontaneous SAH.
Who Masked: Participant, Care Provider
Masking Description: This clinical trial will be double-blind, with participants and investigators unaware of which treatment arm they have been assigned to.
  Blinding will be done automatically by code assignment via the RedCap electronic database. Only the investigating physician can assign the code to the patient and unblind the patient at the same time. The data manager will have a list of codes for possible unblinding.
  Unblinding the patient for any reason is considered a protocol deviation. The reason for unblinding will be described in the source documentation and recorded in the eCRF. In an emergency, the investigator may perform unblinding himself according to ICH GCP E6(R2) paragraph 4.7.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active - Parecoxib (Experimental): Parecoxib 40 mg/100 ml will be injected into a peripheral or central venous catheter within 12 hours of the patient's inclusion in the study (from when informed consent is signed). Parecoxib 40 mg/100 ml is administered every 12 hours for 5 days. The maximum daily dose is 80 mg.
  In patients with moderate hepatic impairment (Child-Pugh score 7-9), parecoxib is started at 20 mg/50 mL and continued at this dose every 12 hours. The maximum daily dose is 40 mg.
  Participants will be monitored for six months for adverse events and changes in subjective status. In the event of adverse events, patients will be followed until resolution. After that, their participation in this clinical trial will be terminated. The total duration of the patient's participation in the clinical trial will be six months.
  Interventions: Drug: Parecoxib
- Control - Placebo (Placebo Comparator): A placebo is a substance administered to a participant as a comparison without any pharmacological effect. However, unlike conventional medicines, it does not contain any active ingredients. In this clinical trial, the placebo is an isotonic sodium chloride solution.
  The placebo is injected into a peripheral or central venous catheter within 12 hours of the patient's enrollment in the study (from when informed consent is signed). Placebo 100 mL per dose will continue to be administered every 12 hours for five days.
  Participants will be followed for six months for any adverse events and changes in subjective status. In the event of adverse effects, patients will be followed until resolution. After that, their participation in this clinical trial will be terminated. The total duration of the patient's participation in the clinical trial will be six months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Parecoxib — Parecoxib (Dynastat) 40 mg solution for injection is for intravenous administration. Parecoxib may be given as an intravenous injection for 30 minutes directly into a vein or through an intravenous infusion set.
  Arms: Active - Parecoxib
Drug: Placebo — Placebo intravenous injection can be administered quickly and directly into a vein or through an intravenous infusion set.
  Arms: Control - Placebo

SUMMARY:
Because of the important role of inflammation in the pathophysiology of SAH, it was hypothesized that its pharmacological manipulation might improve the prognosis of patients. In recent years, the effects of several groups of anti-inflammatory drugs on the development of complications after SAH have been described. Initially promising, glucocorticoids, thought to reduce cerebrovascular inflammation, brain swelling, and headache, failed in clinical trials. Studies have not provided clear evidence of the beneficial effects of these drugs in patients after SAH. Therefore, the administration of glucocorticoids is not currently part of the recommended practice. In addition, glucocorticoid treatment is associated with adverse effects that worsen outcomes, including hyperglycemia, infection, and the risk of gastrointestinal bleeding.

DETAILED DESCRIPTION:
Spontaneous subarachnoid hemorrhage (SAH) is a specific type of hemorrhagic stroke with a worldwide incidence ranging from 0.5 to 28 per 100,000 population, with large regional variations. Despite improvements in diagnosis, treatment and care, SAH remains a disease with high mortality and morbidity. According to the literature, one third of patients die within the first few days after SAH, and most survivors have cognitive impairment or long-term disability. The overall clinical outcome depends on the severity of early brain injury (EBI), cerebral edema, hydrocephalus, development of delayed ischemic neurological deficit (DIND), epileptic seizures, and other complications. The pathophysiological cascades responsible for the development of these complications remain poorly understood. However, numerous studies support the important role of aseptic cerebrovascular inflammation induced by blood and blood breakdown products in the subarachnoid space after SAH. The increased interest in the development of cerebrovascular inflammation after SAH is confirmed by the increasing number of clinical and experimental studies devoted to this topic. Cerebrovascular aseptic inflammation as a potential treatment target is also mentioned in current guidelines for the management of patients after SAH.

The results of experimental studies formed the basis for the clinical evaluation of the effects of NSAIDs after SAH. The effects of several commonly used NSAIDs, particularly dexketoprofen, ibuprofen, diclofenac, indomethacin, or dipyrone, have been evaluated in prospective and retrospective clinical trials over the past decade. In addition to reducing pro-inflammatory markers such as IL6, lowering body temperature and platelet aggregation, the administration of NSAIDs has been associated with reduced mortality and improved clinical outcomes. Despite the beneficial effects of some NSAIDs, more robust studies are still lacking, except for one study that evaluated the effect of meloxicam in patients after SAH. This study was a randomized, double-blind, placebo-controlled trial. It showed a trend towards a better outcome with a lower incidence of vasospasm or mortality in patients after SAH.

Despite encouraging experimental results, no clinical trials have yet evaluated the anti-inflammatory and other potentially beneficial effects of cyclooxygenase-2 (COX-2) inhibitors. COX-2 inhibitors, or coxibs, belong to the group of NSAIDs that selectively inhibit the COX-2 enzyme, which is responsible for developing inflammation and pain. A planned clinical study will evaluate the effects of parecoxib, a specific COX-2 inhibitor in the NSAIDs group, on overall clinical outcome and development of complications in patients following spontaneous SAH.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age: 18-85 years
* Weight> 50 kg
* Spontaneous SAH diagnosed on a native CT brain max. 48 hours after the first symptoms
* Spontaneous SAH caused by rupture of the cerebral aneurysm confirmed on DSA or CT angiography (Fisher grade 1 to 4) OR Spontaneous SAH without a source on CT AG, DSA or MRI with Fisher grade 3 and 4
* For women capable of becoming pregnant (see definitions from the CTFG guideline for contraception): use of the following highly reliable contraceptive method within 3 months after the end of the study: adherence to sexual abstinence or contraception containing progesterone with inhibition of ovulation (oral administration, injection) or non-hormonal intrauterine device or hormonal or bilateral tubal occlusion or partner vasectomy. Males: adherence to sexual abstinence or use of an adequate contraceptive method (i.e. condom) in case of sexual intercourse within 3 months after the end of the study.

Exclusion Criteria:

* Symptoms of SAH without the finding of blood on the initial native CT scan of the brain
* SAH from a cause other than a ruptured aneurysm, e.g. A-V malformation, traumatic SAH
* Pregnancy and breastfeeding (pregnancy test)
* Known hypersensitivity to the components of the product
* Allergic reaction to the active substance or sulfonamides in the anamnesis
* Concomitant treatment with other non-steroidal anti-inflammatory drugs, aspirin or corticosteroids (at least five half-lives before administration of the medicinal product under investigation)
* Severe hepatic insufficiency (serum albumin level <25 g/l or Child-Pugh score less than 10).
* Active peptic ulcer or bleeding from the gastrointestinal tract in the anamnesis
* Inflammatory bowel disease in the anamnesis
* Congestive heart failure (NYHA II-IV) in history.
* Proven ischemic heart disease, peripheral arterial insufficiency.
* Participation in another clinical study (a gap of at least five half-lives before administration of the medicinal product under investigation).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Influence of parecoxib on outcome of patients with SAH | 180 days ± 14 days after first dose of parecoxib/placebo
  The primary outcome measure is the percentage of patients in the active and control groups whose outcome is categorized as favorable (mRS 0-3) or unfavorable (mRS 4-6) according to the modified Rankin Scale (mRS).

SECONDARY OUTCOMES:
Influence of parecoxib on outcome of patients with SAH | Discharge from hospital and 90 days ± 7 days after first dose of parecoxib/placebo
  The secondary monitored parameter is the percentage of patients in the active and control groups whose outcome, according to the modified Rankin scale (mRS), is divided into favourable (mRS 0-3) or unfavourable (mRS 4-6).
Occurrence of symptomatic vasospasms (vasospasms confirmed on TCD / CT AG / MR AG / DSA | Six, eight and ten days after the application of the first dose of the evaluated medicinal product /placebo.
  Number of patients with vasospasms confirmed on TCD / CT AG / MR AG / DSA
Incidence of delayed ischemic neurological deficit (DIND) | Six, eight and ten days, three and six months after the application of the first dose of the evaluated medicinal product /placebo.
  Number of patients with delayed ischemic neurological deficit
Mortality | During the treatment and post treatment period of hospitalization, 90 days ± 7 days and 180 days ± 14 days
  Number of deaths
Length of hospitalization in ICU | 3 months
  Length of hospitalization in ICU
Total length of hospitalization | 3 months
  Total length of hospitalization
Occurrence of acute hydrocephalus | During the treatment and post treatment period of hospitalization
  Number of patients with acute hydrocephalus
Occurrence of chronic hydrocephalus | During the treatment and post treatment period of hospitalization, 90 days ± 7 days, 180 days ± 14 days
  Number of patients with chronic hydrocephalus with V-P shunt implantation
Occurrence of fevers | During the treatment and post treatment period of hospitalization
  Number of patients with fever above 38 degrees Celsius
Occurrence of inflammation | During the treatment and post treatment period of hospitalization
  Evaluation of the systemic inflammatory response (assessed daily during hospitalization) meeting at least 2 parameters:
  * heart rate > 90/min.
  * leukocytosis > 12x109/l) or leukopenia < 9x109
  * respiratory rate > 20/min. or PaCO2 < 32 mm Hg (4.3 kPa)
  * body temperature < 36.0 °C or > 38.0 °C
Evaluation of pain according to Visual Analogue Scale | During the treatment and post treatment period of hospitalization, discharge from hospital, 90 days ± 7 days and 180 days ± 14 days after first dose of parecoxib/placebo
  The comparison of the patients in the treatment and placebo arm with pain according to the Visual Analogue Scale, a numerical scale from 0 to 10 points, where increasing pain is indicated by a higher score.
Evaluation of prostaglandins and pro-inflammatory cytokines in the cerebrospinal fluid in the case of the below-mentioned external ventricular drainage after 2 days and in the serum | 0, 2, 4, 6, 8 and 10 days after implantation of drainage
  Evaluation of prostaglandins (COX-2, PGH2, PGI2, PGE2, PGD2, PF2a, TXA2) and pro-inflammatory cytokines (TNF, IL-1, IL-4, IL-6, IL-8, IL-12) in the cerebrospinal fluid in the case of the below-mentioned external ventricular drainage after 2 days and in the serum regardless of the established cerebrospinal fluid drainage after two days to day 10 from initial symptoms
Evaluatioon of laboratory markers of inflammatory response in peripheral blood | Two, four, six, eight and ten days after the application of the first dose parecoxib/placebo
  C-reactive protein (CRP), procalcitonin (PCT) and white blood cell count
Evaluation of the functionality of the blood-cerebrospinal fluid barrier every 2 days if cerebrospinal fluid drainage is necessary. | 0, 2, 4, 6, 8 and 10 days after implantation of drainage
  This evaluation will compare the number of patients in the treatment and placebo arms who undergo cerebrospinal fluid drainage.
Quality of life measured through questionnaires | Discharge from hospital, 90 days ± 7 days and 180 days ± 14 days after the application of the first dose parecoxib/placebo
  Evaluation of quality of life (SF-36 score)
Evaluation of the difference in efficacy parameters between subgroups according to the source of bleeding | After discharge from hospital, six days after administration of the 1st dose of parecoxib/placebo
  Number of patients with inflamation based on source of bleeding
Serious adverse events | During hospitalization, at discharge, 90 days ± 7 days, 180 days ± 14 days after the first dose of parecoxib/placebo
  Percentage of patients in the experimental and placebo groups with the occurrence of serious adverse events (SAE) (assessed during hospitalization, at discharge, 3 and 6 months after the first dose) supplemented by evaluation in individual subgroups according to the source of bleeding.
Hepatotoxicity | Before the 1st dose of parecoxib/placebo, 1., 3. and 5. day of treatment and 10. day of hospitalization
  Percentage of patients in the experimental and placebo groups with an increase in blood creatine phosphokinase (CPK), an increase in blood lactate dehydrogenase (LDH), an increase in alanine transaminase (ALT), an increase in aspartate transaminase (AST), and an increase in blood urea level > 5x ULN; separate analysis for subgroups by source of bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Solar, Principal Investigator — St. Anne´s University Hospital Brno
Locations (1):
- St. Anne's University Hospital Brno, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No